CLINICAL TRIAL: NCT05293665
Title: A Phase 3 Multi-Center International, Randomized, Active-Controlled Platform Trial to Compare Homologous Boost of Authorized COVID-19 Vaccines and Heterologous Boost With UB-612 Vaccine
Brief Title: Platform Trial to Compare Homologous Boost of Authorized COVID-19 Vaccines and Heterologous Boost With UB-612 Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vaxxinity, Inc. (Industry)
Collaborators: Syneos Health (Other); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UB-612-305; U1111-1276-9528 (Other: WHO); 2022-000088-38 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-24 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Vaccines
Keywords: COVID-19; SARS-CoV-2; peptide; vaccine; subunit; protein
MeSH Terms: conditions — COVID-19 | interventions — UB-612 COVID-19 vaccine; BNT162 Vaccine; BIBP COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Platform trial with multiple sub-studies. Each sub-study has two treatment arms: active comparator and IMP.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- double-blind UB-612 boost of ChAdOx1-S (Experimental): A single injection of UB-612 on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with ChAdOx1-S.
  Interventions: Biological: UB-612
- double-blind ChAdOx1-S boost (Active Comparator): A single injection of ChAdOx1-S on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with ChAdOx1-S.
  Interventions: Biological: ChAdOx1-S vaccine
- double-blind UB-612 boost of BNT162b2 (Experimental): A single injection of UB-612 on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with BNT162b2
  Interventions: Biological: UB-612
- double-blind BNT162b2 boost (Active Comparator): A single injection of BNT162b2 on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with BNT162b2.
  Interventions: Biological: BNT162b2 vaccine
- double-blind UB-612 boost of Sinopharm BIBP (Experimental): A single injection of UB-612 on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with Sinopharm BIBP.
  Interventions: Biological: UB-612
- double-blind Sinopharm BIBP (Active Comparator): A single injection of Sinopharm BIBP on Day 1 in a double-blinded fashion in subjects who completed the primary immunization series with Sinopharm BIBP.
  Interventions: Biological: Sinopharm BIBP
- open-label UB-612 boost of BNT162b2 (Experimental): A single injection of UB-612 on Day 1 in an open-label fashion in subjects who completed the primary immunization series with BNT162b2.
  Interventions: Biological: UB-612
- open-label BNT162b2 boost (Active Comparator): A single injection of BNT162b2 on Day 1 in an open-label fashion in subjects who completed the primary immunization series with BNT162b2.
  Interventions: Biological: BNT162b2 vaccine

INTERVENTIONS:
Biological: UB-612 — UB-612 (100µg), 0.5mL suspension, intramuscular injection
  Arms: double-blind UB-612 boost of BNT162b2; double-blind UB-612 boost of ChAdOx1-S; double-blind UB-612 boost of Sinopharm BIBP; open-label UB-612 boost of BNT162b2
Biological: BNT162b2 vaccine — BNT162b2 vaccine (30µg), 0.3mL suspension, intramuscular injection
  Arms: double-blind BNT162b2 boost; open-label BNT162b2 boost
Biological: ChAdOx1-S vaccine — ChAdOx1-S vaccine, 0.5 mL suspension with approximately 5.0 × 10˄10 viral particles, intramuscular injection
  Arms: double-blind ChAdOx1-S boost
Biological: Sinopharm BIBP — Sinopharm BIBP COVID-19 vaccine, 0.5mL (4µg) suspension, intramuscular injection
  Arms: double-blind Sinopharm BIBP

SUMMARY:
This is a multicenter, international, randomized, active-controlled platform study with each sub-study designed to randomize subjects to receive a single injection with UB-612 or a comparator COVID-19 vaccine in 1:1 ratio.

DETAILED DESCRIPTION:
The current platform protocol is designed to determine the safety and immunizing activity of a booster dose of 100 μg UB-612 in patients who have received a different vaccine 3 months or more before the study start (i.e., Day 1). The randomized, active-controlled multicenter study sponsored by Vaxxinity will be conducted in several countries under a master platform protocol outlining common objectives, endpoints, population, study design, and data analysis. The platform protocol is designed for multiple sub-studies to be implemented at any time, each independently addressing the same set of scientific questions aimed to evaluate the immune responses after a booster injection with UB-612 vaccine candidate and a particular comparator COVID-19 vaccine product.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent/assent after reading the consent/assent form and having adequate opportunity to discuss the study with an investigator or designee.
2. Documented fully vaccinated with primary series of a comparator vaccine. Primary immunization is defined as 2 doses spaced approximately 3-16 weeks apart. The last dose of the previous vaccine must have been administered at least three (3) months (Pfizer at least (5) months) prior to Day 1, taking into consideration the current local and national regulations, and according to details related to individual comparators provided in relevant sub-studies. Documentation, such as the National Health Service (NHS) COVID Pass, United States Centers for Disease Control vaccine card, or equivalent documentation (e.g., medical records, vaccine passport; in accordance with local approved vaccination record documentation) will be required for proof of vaccination, vaccine manufacturer and vaccination dates.
3. No clinically significant health problems that could affect the safety of the subject, as determined by the investigator by medical history, laboratory tests and physical examination. May have a stable pre-existing medical condition that did not require significant change in medication or hospitalization in 3 months before screening or which, in the judgement of the investigator is unlikely to require a significant change in therapy or hospitalization for worsening disease in the 3 months after Day 1.
4. Negative SARS-CoV-2 reverse transcriptase-polymerase chain reaction (RT-PCR) or antigen test within 24-48 hours prior to receipt of injections on Day 1.
5. Female subjects of non-childbearing potential may be enrolled.
6. Males and WOCBP, 16 years or older, may be enrolled in the study if they are willing to practice abstinence from sexual intercourse or are willing to use acceptable methods of contraception as described below, from the time of signing the informed consent/assent during the screening period through study product injection on Day 1 and until completion of Day 29. Acceptable methods of contraception should be consistent with local availability/regulations regarding the use of contraceptive methods for those participating in clinical trials.
7. For WOCBP, a serum or urine pregnancy test must be negative at Screening and on the day of study product injection.
8. Must be able to read, understand, and complete questionnaires and diary entries.
9. Plans to reside within study area for the duration of the study.
10. Able to comply with study procedures for the full duration of the study, in the opinion of the investigator.

Exclusion Criteria:

1. Known history of COVID-19 or SARS-CoV-2 infection within six (6) months prior to vaccination (Day 1).
2. Receipt of a booster COVID-19 vaccination in addition to the primary vaccine series.
3. Presence of fever >100.4°F/38°C or other signs or symptoms of COVID-19 (e.g., chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea) within 1 week prior to Day 1 study product injection. Screening and/or study product injection may be rescheduled at the discretion of the investigator.
4. Clinical manifestations of systemic diseases considered by the investigator to impact safety or immunogenicity.
5. Prior history of pericarditis or myocarditis of any etiology.
6. Prior history of thrombosis of major vessels, including cerebrovascular or splanchnic thrombosis or of thrombosis with thrombocytopenia syndrome
7. History of anaphylaxis (vaccine related or not).
8. Chronic kidney disease with dialysis.
9. Receipt of systemic corticosteroids (≥0.5 mg/kg per day of prednisone or equivalent)for ≥7 days is prohibited from 28 days before enrollment through conclusion of the study. Topical, inhaled, intra-nasal, intra-articular or intra-bursal administration of corticosteroids is permitted.
10. Receipt of any cytotoxic or immunosuppressive drug or biologics six (6) months prior to Day 1 visit.
11. Receipt of any investigational drug within six (6) months prior to Day 1 visit.
12. Subject received or plans to receive a live attenuated vaccine or licensed adjuvanted(non-aluminum compound) vaccination within 28 days before or after planned administration of study vaccine (Day 1) or another type of vaccine (including influenza vaccine) within 14 days prior to or after planned administration of study vaccine on Day1 visit.
13. Human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg) positive; hepatitis C virus (HCV) antibody positive subjects may be tested for RNA and if negative may be enrolled.
14. Any Grade 2 or greater clinical or laboratory abnormalities at screening results.

    Grade 1 abnormal clinical or laboratory adverse event screening test results which, according to the investigator, are non-clinically significant would not disqualify a potential subject. Clinical or laboratory screening tests may be repeated once to exclude transient abnormalities.
15. Immunocompromised state (weakened immune system) from solid organ transplant, immunosuppressive or immunodeficient state, autoimmune diseases, asplenia and, recurrent severe infections.
16. Have an active malignancy or history of metastatic or hematologic malignancy except non-melanoma skin cancers.
17. Pregnant or breastfeeding female, or female who intends to become pregnant during the study period.
18. Administration of immunoglobulins and/or any blood products within the 120 days preceding Day 1 or planned administration during the study period.
19. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
20. Bilateral tattoos or scars at the deltoid sites of intramuscular (IM) injection that would obscure examination of injection site reactions.
21. Behavioral, cognitive, or psychiatric disease that, in the opinion of the Principal Investigator or his or her representative physician, affects the subject's ability to understand and cooperate with all study protocol requirements.
22. Any alcohol or drug abuse over the 12 months prior to enrollment in the study that has caused medical, professional, or family problems, indicated by clinical history.
23. Grade 2 or higher hypertension (systolic >160 mm Hg and/or diastolic >100 mm Hg).
24. Any other condition that, in the opinion of the Principal Investigator or his/her representative physician, could put the safety/rights of potential subjects at risk or prevent them from complying with the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 944 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Presence of solicited local or systemic reactions | Day 8 after injection
  Local: pain, tenderness, erythema, induration, pruritis. Systemic: Nausea, diarrhea, headache, fatigue, myalgia, chills, joint pain, rash
Presence of unsolicited local or systemic reactions | Day 29 after injection
  Any AE reported by the subject that is not specified as a solicited
Presence of serious adverse events | Day 387 after injection
  SAE are reported through the study
Presence of medically attended adverse events | Day 387 after injection
  AE that leads to an unscheduled visit
Presence of adverse events of special interest | Day 387 after injection
  AESI are reported throughout the study
Boost in neutralizing antibody titers against Wuhan strain at Day 29 | Day 29 after injection
  Geometric Mean Titer Ratios of neutralizing antibodies at Day 29 determined using replicating or pseudotyped virus

SECONDARY OUTCOMES:
Boost in neutralizing antibody titers against Omicron strain at Day 29 | Day 29 after injection
  Geometric Mean Titer Ratios of neutralizing antibodies at Day 29 determined using replicating or pseudotyped virus
Responders determined on Day 29 (Wuhan) | Day 1 to 29 after injection
  Proportion of subjects with ≥4-fold antibody titer rise from Day 1 to Day 29
Responders determined on Day 29 (Omicron) | Day 1 to 29 after injection
  Proportion of subjects with ≥4-fold antibody titer rise from Day 1 to Day 29
Kinetics and duration of antibody response - Responders via neutralizing antibodies | Day 1 to Day 15, Day 29, and Months 6 and 12
  Proportion of subjects with ≥4-fold antibody titer rise over the life of trial measured by neutralizing antibodies determined using replicating or pseudotyped virus
Kinetics and duration of antibody response - Responders via binding to S1-RBD | Day 1 to Day 15, Day 29, and Months 6 and 12
  Proportion of subjects with ≥4-fold antibody titer rise over the life of trial measured by IgG antibodies titers measured by direct S1-RBD binding ELISA
Kinetics and duration of antibody response - GMFI via neutralizing antibodies | Day 1 to Day 15, Day 29, and Months 6 and 12
  Geometric Mean Fold Increase of neutralizing antibodies determined using replicating or pseudotyped virus
Kinetics and duration of antibody response - GMFI via binding to S1-RBD | Day 1 to Day 15, Day 29, and Months 6 and 12
  Geometric Mean Fold Increase of IgG antibodies titers measured by direct S1-RBD binding ELISA
Kinetics and duration of antibody response - AUC via neutralizing antibodies | Day 15 to Month 12
  Area under the curve (AUC) by treatment group and virus variants calculated from neutralizing antibody response determined using replicating or pseudotyped virus
Kinetics and duration of antibody response - AUC via binding to S1-RBD | Day 15 to Month 12
  Area under the curve (AUC) by treatment group and virus variants calculated from IgG antibody response measured by direct S1-RBD binding ELISA
Kinetics and duration of antibody response - GMT via neutralizing antibodies | Days 15, 29, and Months 6 and 12
  Geometric Mean Titers measured by neutralizing antibody response by treatment group and virus variants
Kinetics and duration of antibody response - GMT via binding to S1-RBD | Days 15, 29, and Months 6 and 12
  Geometric Mean Titers measured by IgG antibody response measured by direct S1-RBD binding ELISA
Kinetics and duration of antibody response - Reverse Cumulative Distribution Curve via neutralizing antibodies | Day 29 and Month 6 and 12
  Distribution of neutralizing antibody titers displayed as reverse cumulative distribution curves by treatment group and virus variants measured by neutralizing antibody response
Kinetics and duration of antibody response - Reverse Cumulative Distribution Curve via binding to S1-RBD | Day 29 and Month 6 and 12
  Distribution of IgG antibody titers displayed as reverse cumulative distribution curves by the treatment group and virus variant measured IgG antibody response measured by direct S1-RBD binding ELISA

OTHER OUTCOMES:
Ability to boost cellular immunity | Days 1, 15 and 29, and Months 6 and 12
  Cytokine secreting spots per million cells and % cells staining for cytokines measured by ELISpot and ICS
Ability to boost humoral immunity (non-neutralizing) | Day 1 and Day 29
  Fc-mediated antibody ADCP (antibody dependent cell-mediated phagocytosis) responses
Ability to boost humoral immunity (neutralizing) against additional variant - GMT via neutralizing antibodies | Day 1 and Day 29
  Geometric Mean Titers in neutralizing antibody titers measured using additional variant replicating or pseudotyped viruses
Ability to boost humoral immunity (neutralizing) against additional variant - GMR via neutralizing antibodies | Day 1 and Day 29
  Geometric Mean Titer Ratios in neutralizing antibody titers measured using additional variant replicating or pseudotyped viruses
Ability to boost humoral immunity (neutralizing) against additional variant - GMFI via neutralizing antibodies | Day 1 and Day 29
  Geometric Mean Fold Increase in neutralizing antibody titers measured additional variant replicating or pseudotyped viruses

CONTACTS AND LOCATIONS:
Locations (7):
- PanAmerican Clinical Research, Brownsville, Texas, United States
- Panama (3):
  - Cevaxin David, David
  - Cevaxin 24 de Dieciembre, Panama City
  - Cevaxin The Panama Clinic, Panama City
- Philippines (3):
  - Health Index Multispecialty, Bacoor
  - Iloilo Doctors Hospital, Iloilo City
  - St Pauls Hospital Iloilo City, Iloilo City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flaxman A, Marchevsky NG, Jenkin D, Aboagye J, Aley PK, Angus B, Belij-Rammerstorfer S, Bibi S, Bittaye M, Cappuccini F, Cicconi P, Clutterbuck EA, Davies S, Dejnirattisai W, Dold C, Ewer KJ, Folegatti PM, Fowler J, Hill AVS, Kerridge S, Minassian AM, Mongkolsapaya J, Mujadidi YF, Plested E, Ramasamy MN, Robinson H, Sanders H, Sheehan E, Smith H, Snape MD, Song R, Woods D, Screaton G, Gilbert SC, Voysey M, Pollard AJ, Lambe T; Oxford COVID Vaccine Trial group. Reactogenicity and immunogenicity after a late second dose or a third dose of ChAdOx1 nCoV-19 in the UK: a substudy of two randomised controlled trials (COV001 and COV002). Lancet. 2021 Sep 11;398(10304):981-990. doi: 10.1016/S0140-6736(21)01699-8. Epub 2021 Sep 1. PMID 34480858
- [Background] Kanokudom S, Assawakosri S, Suntronwong N, Auphimai C, Nilyanimit P, Vichaiwattana P, Thongmee T, Yorsaeng R, Srimuan D, Thatsanatorn T, Klinfueng S, Sudhinaraset N, Wanlapakorn N, Honsawek S, Poovorawan Y. Safety and Immunogenicity of the Third Booster Dose with Inactivated, Viral Vector, and mRNA COVID-19 Vaccines in Fully Immunized Healthy Adults with Inactivated Vaccine. Vaccines (Basel). 2022 Jan 6;10(1):86. doi: 10.3390/vaccines10010086. PMID 35062747
- [Background] Petrosillo N, Viceconte G, Ergonul O, Ippolito G, Petersen E. COVID-19, SARS and MERS: are they closely related? Clin Microbiol Infect. 2020 Jun;26(6):729-734. doi: 10.1016/j.cmi.2020.03.026. Epub 2020 Mar 28. PMID 32234451
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Matthes H, Herbst H, Schuppan D, Stallmach A, Milani S, Stein H, Riecken EO. [Distribution of procollagen transcripts in chronic inflammatory bowel diseases using in situ hybridization]. Verh Dtsch Ges Inn Med. 1991;97:12-7. No abstract available. German. PMID 1808876
- [Derived] Rumyantsev A, Wang L, Wang S, Kemp T, Wriggins A, Burks A, Fisher D, Brokke K, Fix A, Hensley S, Lewis M, Zhu R, Wang K, Shasha C, Piccini G, Manenti A, Montomoli E, DeAntonio R, Saez-Llorens X, Chan M, Alberto E, Lallaine Borra MD, Jaen AM, Heppner G, Palm U, Monath TP. Safety and immunogenicity of UB-612 heterologous booster in adults primed with mRNA, adenovirus, or inactivated COVID-19 vaccines: a randomized, active-controlled, Phase 3 trial. EClinicalMedicine. 2025 Jul 21;86:103349. doi: 10.1016/j.eclinm.2025.103349. eCollection 2025 Aug. PMID 40727012
- [Derived] Wang CY, Peng WJ, Kuo BS, Ho YH, Wang MS, Yang YT, Chang PY, Shen YH, Hwang KP. Toward a pan-SARS-CoV-2 vaccine targeting conserved epitopes on spike and non-spike proteins for potent, broad and durable immune responses. PLoS Pathog. 2023 Apr 20;19(4):e1010870. doi: 10.1371/journal.ppat.1010870. eCollection 2023 Apr. PMID 37079651
- See also: Vaxxinity Homepage — https://vaxxinity.com/